CLINICAL TRIAL: NCT06208839
Title: 1R44DA050214 - 01 Mobile Technologies Extending Reach of Primary Care for Substance Use
Brief Title: Mobile Technologies Extending Reach of Primary Care for Substance Use Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chess Mobile Health (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Western Michigan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2023-SBIR-ChessHealth; 1R44DA050214-01 (NIH)
Record Dates: First submitted 2023-12-14; First posted 2024-01-17 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Substance-Related Disorders
Keywords: Substance Use Disorder; Screening, Brief Intervention, Referral, and Treatment
MeSH Terms: conditions — Substance-Related Disorders | interventions — Ethanol; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SBIRT/TAU for those with moderate risk drug or alcohol use (Active Comparator): This moderate risk group will receive the standard Screening and Brief Intervention Treatment (SBIRT) along with Treatment as Usual (TAU) at the clinic.
  Interventions: Other: SBIRT/TAU for those with moderate risk drug or alcohol use
- SBIRT/eIntervention for those with moderate risk drug or alcohol use (Experimental): Subjects assigned to this condition will be instructed by the research assistant in how to download and use the eIntervention app, which they will be free to use as they like for the duration of the study. The app will contain a personalized suite of programs and activities. Unlike the TAU condition, the patient's referral to treatment would be managed through eIntervention. For example, the app will show the patient their referral details (if a referral to treatment was made), including details on the provider, referred services, and contact information, and will offer them videos of peers and professionals educating them on addiction, treatment, and sharing personal stories of recovery.
  Interventions: Device: SBIRT/eIntervention for those with moderate risk drug or alcohol use
- SBIRT/TAU for those assessed with high risk. (Active Comparator): This high risk group will receive the standard Screening and Brief Intervention Treatment (SBIRT) along with Treatment as Usual (TAU) at the clinic.
  Interventions: Other: SBIRT/TAU for those assessed with high risk.
- SBIRT/eIntervention those assessed with high risk. (Experimental): Subjects assigned to this condition will be instructed by the research assistant in how to download and use the eIntervention app, which they will be free to use as they like for the duration of the study. The app will contain a personalized suite of programs and activities. Unlike the TAU condition, the patient's referral to treatment would be managed through eIntervention. For example, the app will show the patient their referral details (if a referral to treatment was made), including details on the provider, referred services, and contact information, and will offer them videos of peers and professionals educating them on addiction, treatment, and sharing personal stories of recovery.
  Interventions: Device: SBIRT/eIntervention those assessed with high risk.

INTERVENTIONS:
Device: SBIRT/eIntervention for those with moderate risk drug or alcohol use — The Connections App is available on iOS or Android and will be offered to the patient during the referral process and contains the following functionalities:
  * Online view of the referrals made for them e.g. to healthcare provider
  * Secure messaging with the referring provider
  * Secure messaging with the destination provider(s) to support them to adhere to the referral, and/or the patient can seek assistance with the destination provider,
  * Informative multimedia content filtered from a library to fit the patient including testimonial content from peers thus showing the patient that others like them have shared their addiction experience and successfully received treatment and achieved recovery,
  * Capture structured feedback from the patient
  The patient may access more functionality within the Connections App for those who wish to modify behavior using eTherapy and eRecovery. eRecovery includes ecological momentary assessments (EMA) selected by the provider.
  Arms: SBIRT/eIntervention for those with moderate risk drug or alcohol use
Device: SBIRT/eIntervention those assessed with high risk. — The Connections App is available on iOS or Android and will be offered to the patient during the referral process and contains the following functionalities:
  * Online view of the referrals made for them e.g. to healthcare provider
  * Secure messaging with the referring provider
  * Secure messaging with the destination provider(s) to support them to adhere to the referral, and/or the patient can seek assistance with the destination provider,
  * Informative multimedia content filtered from a library to fit the patient including testimonial content from peers thus showing the patient that others like them have shared their addiction experience and successfully received treatment and achieved recovery,
  * Capture structured feedback from the patient
  The patient may access more functionality within the Connections App for those who wish to modify behavior using eTherapy and eRecovery. eRecovery includes ecological momentary assessments (EMA) selected by the provider.
  Arms: SBIRT/eIntervention those assessed with high risk.
Other: SBIRT/TAU for those with moderate risk drug or alcohol use — Treatment as usual
  Other Names: Treatment as usual group[
  Arms: SBIRT/TAU for those with moderate risk drug or alcohol use
Other: SBIRT/TAU for those assessed with high risk. — Treatment as usual for high risk group
  Other Names: High risk treatment as usual
  Arms: SBIRT/TAU for those assessed with high risk.

SUMMARY:
The goal of this clinical trial is to evaluate efficacy of our enhanced version of the CHESS Health eIntervention in a clinical setting for those with moderate risk drug or alcohol use and those at high risk or with Substance Use Disorder (SUD) as measured by the ASSIST and the AUDIT assessment tools. The clinical trial is designed to determine whether SBIRT/eIntervention is significantly more effective than SBIRT/Treatment as usual (TAU) as delivered in a primary care setting. While it is not feasible or practical to individually test all components and features of the planned eIntervention, this design will permit testing of efficacy for reduction of substance use in both risk groups and increased enrollment in treatment for the high risk/SUD group in the SBIRT/eIntervention cohorts compared to the SBIRT/TAU cohorts. Note that the investigators are not including a screening/assessment only or other control condition, as the purpose of this clinical trial is not to test the efficacy of SBIRT itself, but rather to test whether SBIRT/eIntervention improves outcomes and successful referral relative to SBIRT/TAU delivery alone.

DETAILED DESCRIPTION:
The investigators will recruit and randomize 200 individuals screening positive on the NIDA Quick Screen.

All participants will receive SBIRT as currently implemented at Western Michigan and as described above. Adult patients would be asked prior to appointments at Western Michigan, either in-person when in a waiting room and/or via email for virtual appointments if they'd would be willing to answer a brief, anonymous online survey regarding their substance use as part of a research study. Upon completing the survey, the results of the survey would be displayed for the patient to see. If the patient's answers to the screening tool indicate their use may be risky or indicates a serious problem regarding assessment, then they would be asked if they would consider participating in a research study (the investigators would provide an online description of the requirements of the study and the payments for participation). If they click through as being interested, the investigators will display more detail about the research study, explain that they will need to review and sign a consent form, and would be required to speak with a research assistant in the coming days. The investigators would present them an electronic consent form and require them to scroll through and, if necessary, could ask them a question or two to confirm their understanding, before allowing them to electronically sign the consent. The investigators would advise them that their participation will not be anonymous. If the patient consents, then the investigators would have them to complete the longer NIDA ASSIST or AUDIT screening tool. If the patient's answers indicate a risk score in the low-risk range for either alcohol or illicit drugs, the investigators will exclude them from continuing in the study.

If the patient's answers indicate a risk score in the moderate to high range, then they would be randomized to the intervention group or the control group. As part of the randomization process, the SBIRT/TAU and the SBIRT/eIntervention groups will have two sub-groups each: (1) those with moderate risk drug or alcohol use and those at high risk or with SUD as measured by the ASSIST and the AUDIT assessment tools). Thus, participants will have been randomized into four cohorts of about 50 subjects each.

If the patient is randomized to the intervention group, then they would be presented a set of digital interventions for them to access then as well as to have access to in the coming weeks/months. If the patient is randomized to the control group, they will receive a 'brief intervention' based on the "Drinker's Checkup" licensed by CHESS Health from San Diego State University.

Whether in the intervention group or the control group, they would be recommended for a referral to treatment. If they're already in SUD treatment, then will exclude them from continuing in the study. If the patient is randomized to the intervention group, then in addition to the referral, they would be given use of the Envoy App with referral details and a TBD set of digital interventions for them to access then as well as to have access to in the coming weeks/months. If the patient is randomized to the control group, then they would only get the referral to treatment plus a basic version of the app that consists solely of the survey engine used for primary data collection. The investigators will conduct a 3-month randomized clinical trial, with a 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18 or over
* receiving primary care at Western Michigan
* identified as having a substance-specific NIDA Modified Assist score of 27 or greater.

Exclusion Criteria:

* non-English speaking
* cannot read at a 3rd grade level,
* have current participation in addiction treatment
* determined to be psychiatrically or medically unstable such that completion of the trial is unlikely.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
NIDA Quick Screen | Screening
  The NIDA Quick Screen is a validated instrument designed to assist providers in screening adults for substance use. The screen simply inquires whether a participant has used drugs (mood-altering, illegal, or prescription for nonmedical reasons), alcohol, or tobacco products within the past year and how often these substances have been used.
The Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) | Screening, 3-month, and 6-month
  The Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) was developed for the World Health Organization (WHO) by an international group of researchers and clinicians as a technical tool to assist with early identification of substance use related health risks and substance use disorders in primary health care, general medical care and other settings
The Alcohol Use Disorders Identification Test (AUDIT) | Screening, 3-month, and 6-month
  The Alcohol Use Disorders Identification Test (AUDIT) is a 10-item screening tool developed by the World Health Organization (WHO) to assess alcohol consumption, drinking behaviors, and alcohol-related problems. We will also administer the AUDIT for patients who screen positive for alcohol via the NIDA Quick Screen.
Demographics | Baseline
  Participant Age
Demographics | Baseline
  Participant Race (American Indian or Alaska Native, Asian, Black or African American, Native Hawaiian or Other Pacific Islander, and White)
Demographics | Baseline
  Participant Biological Sex (Male/Female)
Demographics | Baseline
  Participant Ethnicity (Hispanic/Latino vs. non-Hispanic/Latino)
TimeLine Follow-back method | Baseline, 3-month, and 6-month
  Self-reports are collected using the TimeLine Follow-back method, a widely used and well-validated technique for collecting information on all types of substance use on a day-by day basis for the full period of each participants trial involvement (covering the 3 months prior to baseline through the end of the follow-up).
Healthcare utilization | Baseline, 3-month, and 6-month
  Self reported treatment utilization (including emergency department visits, hospitalization, specialty care visits, attendance at self-help meetings) in all conditions.
Contemplation ladder | Baseline, 3-month, and 6-month
  To assess patient motivation
Satisfaction survey | 3-month, 6 month
  Evaluate patients' satisfaction with treatment and interventions

CONTACTS AND LOCATIONS:
Overall Officials: Hans Morefield, Principal Investigator — CHESS Health
Locations (1):
- WMed Health Family Medicine, Kalamazoo, Michigan, United States